CLINICAL TRIAL: NCT04520633
Title: Measurement Properties Validity of the French Traduction of the Severe Asthma Questionnaire: a Prospective Study
Brief Title: Validity of a French Version of the Severe Asthma Questionnaire
Acronym: TRAQUE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200818; 2020-AO1394-35 (Other: IDRCB)
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Asthma
Keywords: severe asthma; quality of life questionnaire
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control level stable: severe asthma for which the control level is stable (variation in ACT score <3 between M0 and M6) contributing to the test-retest
- biologic initiation: introduction or modification of biotherapy at M0
  Interventions: Other: biologic initiation

INTERVENTIONS:
Other: biologic initiation — introduction or modification of biotherapy at M0
  Groups: biologic initiation

SUMMARY:
"Severe asthma affects only 5% of asthmatics, but has a considerable impact on patients owing to the respiratory disability linked to asthma but also complications from oral corticosteroid (OCS) therapy.

Biologics have recently been made available, and improve quality of life (QoL)severe asthma patients. Having a reproducible and reliable measuring tool of QoL for severe asthmatics would be useful for assessing the impact of the various interventions proposed.

QoL questionnaires currently used in respiratory diseases are not specific to severe asthma. They are very focused on respiratory disability, but for example do not take into account the impact of treatments, especially oral steroids.

The Severe Asthma Questionnaire (SAQ) is the very first tool specifically designed to assess the health related quality of life of severe asthma population. The development of its use goes through the validation of this questionnaire in its French translation available since September 2019. "

DETAILED DESCRIPTION:
"Difficult to treat asthma affects about 17% of the asthma population, among which 5% have severe asthma.

For these patients, the disease is often a burden to their professional, family and personal life, significantly altering their quality of life.

Current recommendations on medical management aim at asthma control and reduction of exacerbations. While there are now biologics that effectively address these objectives, they are still struggling to demonstrate their effectiveness in term of quality of life improvement.

Although in real life, patients well responding to biologics often report ""a changing life"", this is not well demonstrated in clinical trials, which only bring out modest variations in quality of life (mainly AQLQ) and asthma control scores. This may be due to the fact that currently used scores, measure either the quality of life in a generic way, or asthma control (dyspnea, use of rescue treatments) rather than asthma specific quality of life, and do not take into account the burden of oral steroids.

For this specific population of asthmatics, even the dedicated scores (11 scales in the adult population and 6 in the pediatric population) have trouble measuring variations in quality of life. They hardly ever manage to demonstrate a difference in quality of life between mild asthma and severe asthma.

However, just like oral steroids sparing, improving quality of life is of concern for physicians.

The development of Patient Reported Outcome (PRO) instruments follows rigorous scientific methodology. The Severe Asthma Questionnaire (SAQ) is a specific instrument for measuring quality of life in severe asthma. It was developed and validated in English by the University of Plymouth in 2018, according to the current recommendations, in an attempt to respond to the lack of specificity of the former quality of life tests.

It has gone through forward and backward translation process into French thanks to the Mappy Trust organization. It seems important to validate, in its French translation, the psychometric properties of the SAQ questionnaire, a specific instrument measuring quality of life for severe asthmatics.

Practical considerations:

* Useful data cf primary and secondary objectives will be collected at the first and the 6th month.
* Standard Operating Procedures: Patient recruitment will only take place in Bichat Hospital. Questionnaires and forms will be lend to the severe asthmatics coming to consultation and day hospital thanks to clinical research associate. Data will be anonymized and collected by a clinical research associate (fulfilled forms and questionnaire and medical file). Data management, data analysis will be ensured by Clinical Research Unit of Bichat Hospital.
* Sample size assessment : estimated on FALISSARD assumption: 320 patients.
* Plan for missing data: usual way for each quality of life questionnaire, enlarged 6th month visit period to collect 6th month reevaluation.
* Statistical analysis plan: cf section primary and secondary objectives.
* Quality assurance plan: Data validation and registry procedures, including any plans for site monitoring and auditing will be ensured by the Clinical Research Unit of Bichat Hospital.
* Data checks: Predefined rules for range will be pre-configure in the eCase Report Form (CRF) computed in REDCap. The data dictionary that contains detailed descriptions of each variable used by the registry (cf inclusion/exclusion criteria, primary and secondary outcome), including the source of the variable, and normal ranges is described in a specific document based on which the eCRF will be built. "

ELIGIBILITY:
Inclusion criteria :

* Adult patients
* Patients diagnosed with severe asthma as defined by the international consensus statement from European Respiratory Society and American Thoracic Society 2014: Asthma which requires treatment for GINA steps 4-5 asthma (high dose Inhaled Cortico Steroids > 1000 micrograms and Long Action Beta Agonist or leukotriene or theophyllin modifier ) for the previous year

  *or systemic CorticoSteroids for 50% of the previous year to prevent it from becoming ''uncontrolled'' or which remains ''uncontrolled'' despite this therapy
* Patient informed and not opposed to participating

Exclusion criteria :

* Lung cancer, heart failure or Chronic Obstructive Pulmonary Disease, or other respiratory disease that may affect the evaluation of asthma
* Patient unable to read French
* Patient unwilling to take part in the research
* Patient under guardianship / curators
* Patient under AME

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe asthma
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Factorial validity of french traduction of SAQ (Severe Asthma Questionnaire ) | 1 month
  Factorial validity (evidence that the instrument measures a single concept): principal component analysis of all items
Internal consistency of french traduction of SAQ | 1 month
  Internal consistency (intercorrelation of items that contribute to a score): Item total correlation and Cronbach's alpha coefficient
Construct validity of french traduction of SAQ | 1 month
  Construct validity (strength of correlation testing a priori hypotheses (discriminant and convergent validity) and degree to which the PRO instrument can distinguish among groups hypothesized a priori to be different (known groups validity)): Spearman correlation between SAQ and ACT*, ACQ*, miniAQLQ*, SGRQ*, SF36*, EQ 5D 5L*, EQ 5D VAS*, OCS dose, Forced expiratory volume in 1s (FEV1))
  * ACT: Asthma Control Test i
  * ACQ: Asthma Control Questionnaire
  * MiniAQLQ: Mini Asthma Quality of Life Questionnaire
  * SGRQ: Saint Georges Respiratory Questionnaire
  * SF36: 36-item Short-Form Health Survey
  * EQ 5D 5L: 5Level-EuroQualityoflife Instrument 5 Dimension
  * EQ 5D VAS: EuroQol Visual Analogue Scale

SECONDARY OUTCOMES:
Usability testing | 6 months
  Questionnaire feasibility: Average filling percentage, mean filling time, need for help in responding, identification of problematic items, reason why they are problematic
Test-retest reliability | 6 months
  Test-retest reliability (stability of scores over time when no change is expected in the concept of interest): intraclass correlation coefficient of SAQ M1 vs M6 within stable ACT score group adjusted on oral corticosteroids dose.
Ability to detect change | 6 months
  Ability to detect change (evidence that a Patient Reported Outcome instrument can identify differences in scores over time in individuals or groups who have changed with respect to the measurement concept): Wilcoxon signed rank-test on oral corticosteroid dose, comparing individuals at M1 and M6 for whom an asthma biotherapy has been initiated in that time interval.
Minimal Clinically Important Difference (MCID) | 6 months
  MCID (minimal difference of significance among any differences observed): anchored base estimation using a global 15point scale ranging scale to measure change.

CONTACTS AND LOCATIONS:
Overall Officials: Camille Taillé, MD-PHD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Bichat-Claude Bernard University Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided